CLINICAL TRIAL: NCT03037502
Title: Tailoring a Lifestyle Intervention to Address Obesity Disparities Among Men
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Collaborators: University of Miami (Other); Vanderbilt University Medical Center (Other); Meharry Medical College (Other); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Derek Griffith, Director of the Center for Research on Men's Health, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 160108; 1U54MD010722 (NIH); NCT04040335 (obsolete NCT alias)
Record Dates: First submitted 2017-01-26; First posted 2017-01-31 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Weight Loss; Obesity
Keywords: Men's Health; weight loss; African American men; Latino men
MeSH Terms: conditions — Weight Loss; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: Tailor Made (Experimental): Intervention Arm: In the pilot intervention, participants will receive: tailored goals/ messages, self-monitoring, weekly small groups to receive health education and community-based information and resources. Participants will also complete two assessment with blood work and anthropometric measurements. These intervention components were selected based on investigator's formative research and experience using them in prior studies. These components will be implemented simultaneously as they complement one another. While all of these components have not been tested together in an intervention for this population, they are variations and enhancements of previous interventions by the investigators.
  Interventions: Behavioral: Tailor Made: Solutions for your health (A su Medida: Soluciones para su salud)
- Comparison (No Intervention): Comparison Condition: Participants in the attention control group will receive self-help materials on how to improve healthy eating, physical activity and weight loss, self-monitoring, and complete two assessments with blood work and anthropometric measurements. Participants in this condition will receive a copy of their assessment data and the nurses will provide this personalized information as well as answer any questions participants may have about their assessment results.

INTERVENTIONS:
Behavioral: Tailor Made: Solutions for your health (A su Medida: Soluciones para su salud) — Assess the effectiveness of a person-specific, randomized controlled pilot weight loss study of 80 African American and 40 Latino men; to compare changes in chronic disease risk behaviors (e.g., diet and physical activity), adiposity measures (e.g., body fat), and psychosocial mediators (e.g., social support, autonomous motivation) between data collected at baseline and at 3-months.
  Arms: Intervention: Tailor Made

SUMMARY:
If the investigators are to adequately address the health needs of African American and Latino men, both culture and gender must be considered when developing and implementing strategies to encourage weight loss and increase their healthy eating and physical activity.The aim of this project is to develop and test gendered, culturally and contextually relevant messages that will be used in a future, web- based tailored intervention to encourage healthy eating and physical activity in African American and Latino men. This study is part of a larger research agenda that for a decade has focused on understanding and reducing chronic disease risk among African American and Latino men. Because men are more likely than women to engage in over 30 behaviors known to increase their risk of injury, morbidity, and mortality, improving men's health requires understanding the social and cultural factors that help explain sex differences in health. Operationalizing gender in individually-tailored health communications has great potential to unlock the potential of health communications and interventions to engage and improve the health of men and particularly African American and Latino men. To date, no community-based intervention has produced clinically significant improvements in weight loss, healthy eating or physical activity in Latino and African American men. It also is unclear how technology can be used to promote these behaviors in this population. Thus, there is a need to develop healthy eating, physical activity and weight loss interventions specifically targeted and tailored to African American and Latino men that explores the utility of technology. This intervention content and focus represents a novel strategy to promote health equity by using technology-based health care innovations to improve healthy eating and active living by addressing a root cause of unhealthy behavior in men: notions of manhood. The investigators focus on gender and manhood because they are under-explored factors that shape men's health behaviors.

DETAILED DESCRIPTION:
The overall aim of this study is to develop and pilot an individualized weight-loss intervention for obese middle-aged African American and Latino men and to explore how the genetically predicted BMI relates to outcomes. Using strategies previously employed by the PI to develop individually-tailored materials for African American men, the proposed study is designed to develop person-specific materials for Latino men (Specific Aim 1). Investigators also will pilot a behavioral weight loss intervention for 35-64 year old African American men in Nashville and Latino men in Miami (Specific Aims 2-3), and explore how the phenotypic expression of obesity shapes and is affected by behavioral and physiological changes (Specific Aim 4). The proposed intervention includes (a) person-specific goals/ messages (via web and text), (b) self-monitoring (via wearable device and text), (c) small group training and education (including social support) and (d) educational and community-based information and resources (via web and text).

ELIGIBILITY:
Inclusion Criteria:

* Age: 35-64 at enrollment
* Race/ ethnicity: African American/ Black or Latino/ Hispanic
* BMI: 27-50
* Fluent in English (Nashville and Miami) or Spanish (Miami)
* Provide informed consent
* Weight less than 400 pounds

Exclusion Criteria:

* Preexisting condition that prohibits at least moderate physical activity
* Serious medical condition that is likely to hinder accurate measurement of weight, for which weight loss is contraindicated or that would cause weight loss
* Prior or planned bariatric surgery
* Chronic use of medications that are likely to cause weight gain or cause weight loss
* No cell phone or land-line phone
* Participant in another obesity, eating or physical activity program or study
* Psychiatric hospitalization or in-patient substance abuse treatment in the last 12 months

Ages: 35 Years to 64 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — This study is interested in piloting a tailored health promoting intervention for African American and Latino men. Thus, recruitment will be open to individuals who self-identify as African American or Latino men, ages 35-64 at enrollment.
Enrollment: 72 (Actual)
Dates: Start 2019-06-12 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-03-31 (Actual)

PRIMARY OUTCOMES:
Change in weight at 3-months post-baseline | 3-months post-baseline of participation
  Investigators will report weight change in absolute terms from baseline.

SECONDARY OUTCOMES:
Percent change in weight at 3-months post-baseline | 3-months post-baseline of participation
  Investigators will report weight change as percent change from baseline.
Change in weight classification | 3-months post baseline of participation
  Investigators will assess change in percentage of participants that regress from obese to overweight classification using BMI in kg/m^2.

OTHER OUTCOMES:
Change in eating practices measured by the Food, Attitudes, and Behaviors Survey (FAB) | 3-months post baseline of participation
  As measured by a modified version of the National Cancer Institute (NCI) 2007 Food Attitudes and Behaviors Survey, to measure the change in fruit and vegetable intake (FVI) during the past month. Responses will be converted into servings, as defined by the MyPyramid 1992 dietary guidelines. Total FVI was calculated as the sum of all items on the screener, excluding fried potatoes.
Change in physical activity measured by the Global Physical Activity Questionnaire (GPAQ) | 3-months post baseline of participation
  The GPAQ measures time spent in vigorous and moderate intensity physical activity. A higher score equates to more physical activity. The range is from 0 - 150 minutes per week.

CONTACTS AND LOCATIONS:
Overall Officials: Emily C Jaeger, MPH, Study Director — Vanderbilt University; Derek M Griffith, PhD, Principal Investigator — Vanderbilt University; Natasha Solle, PhD, Principal Investigator — University of Miami; Neysari Arana, MPH, Study Director — University of Miami
Locations (2):
- United States (2):
  - University of Miami, Miami, Florida
  - Vanderbilt University, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Griffith DM, Jaeger EC, Valdez LA, Schaefer Solle N, Garcia DO, Alexander LR. Developing a "Tailor-Made" Precision Lifestyle Medicine Intervention for Weight Control among Middle-aged Latino Men. Ethn Dis. 2020 Apr 2;30(Suppl 1):203-210. doi: 10.18865/ed.30.S1.203. eCollection 2020. PMID 32269462

DOCUMENTS (1):
  • Informed Consent Form (2019-12-16): https://cdn.clinicaltrials.gov/large-docs/02/NCT03037502/ICF_000.pdf